CLINICAL TRIAL: NCT02377089
Title: Neuromodulation as a New Treatment for Post-Traumatic Stress Disorder in Veterans: Evaluating the Effectiveness of Trigeminal Nerve Stimulation
Brief Title: Neuromodulation for Post-Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: VA Greater Los Angeles Healthcare System (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Andrew F. Leuchter, Professor of Psychiatry and Biobehavioral Sciences, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: W81XWH-14-2-0125
Record Dates: First submitted 2014-11-17; First posted 2015-03-03 (Estimated); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Trigeminal Nerve Stimulation; Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham (Sham Comparator): The stimulators are the same device for the active and sham treatment conditions.
  Interventions: Device: Placebo
- Active (Active Comparator): The stimulators are the same device for the active and sham treatment conditions.
  Interventions: Device: Trigeminal Nerve Stimulation

INTERVENTIONS:
Device: Trigeminal Nerve Stimulation — Subjects will be randomized to treatment with either active or sham TNS for a period of eight weeks. The programming will be set by an individual who has no contact with subjects to deliver TNS in a double-blind manner (n=37 in each group) at the active frequency of 120 Hz. TNS will be performed for approximately 8 hours each night, a protocol that subjects found acceptable in the pilot work.
  Other Names: TNS
  Arms: Active
Device: Placebo — Subjects will be randomized to treatment with either active or sham TNS for a period of eight weeks. The programming will be set by an individual who has no contact with subjects to deliver TNS in a double-blind manner (n=37 in each group) at the sham frequency of 0 Hz. TNS will be performed for approximately 8 hours each night, a protocol that subjects found acceptable in the pilot work.
  Arms: Sham

SUMMARY:
The investigators propose to use a clinical trial to test Trigeminal Nerve Stimulation (TNS) to examine the efficacy of TNS as a new treatment for Post Traumatic Stress Disorder (PTSD) in veterans. Recruitment will take place at the PTSD Outpatient Clinic at the Veterans Affair Greater Los Angeles (VA GLA). Study participants will be asked to complete, at most, 9 assessments/questionnaires regarding their PTSD symptoms and quality of life, use the TNS device every night for 8 hours, log their use of the device, and attend weekly visits to monitor safety and complete assessments. Each subject will be asked to attend 8 visits over the course of 8 weeks. Subjects who receives the sham-controlled treatment will have an additional follow-up phone visit 4 weeks after the week 8 endpoint to examine symptom improvements.

Enrollment and subject-related procedures are projected to take approximately 36 months. Preparations for clinical trial, clinical trial/study procedures and data analysis will occupy a 6 month period, a 36 month period, and a 6 month period, respectively. The duration of this project is approximately 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. 21-65 years old and be a patient in the Post Traumatic Stress Disorder(PTSD) Clinic at the Veterans Affair Greater Los Angeles
2. have experienced trauma while serving in a war zone in Iraq or Afghanistan
3. meet The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria for current war zone-related PTSD with a duration of at least 3 months
4. have completed a course of Prolonged Exposure(PE) therapy in the Resident Psychotherapy Program in the PTSD Clinic within six months of enrollment and with significant residual PTSD symptoms as evidenced by a Clinician-Administered PTSD Scale score >50
5. consent to be randomized to active or sham Trigeminal Nerve Stimulation treatment
6. if receiving medication for depression, anxiety, sleep, or mood stabilization, must have been on stable dose for at least six weeks prior to randomization.

Exclusion Criteria:

1. current substance abuse not in remission for at least 3 months
2. a history of bipolar, schizophrenia, other psychotic disorder, or dementia
3. current suicidal or homicidal ideation requiring hospitalization, or suicide attempt within six months
4. report of severe Traumatic Brain Injury (TBI) with coma duration (30 minutes or more) during the screening interview and/or duration of post - traumatic amnesia (1hour or greater) on the Post-traumatic Amnesia Questionnaire (PTAQ)
5. evidence of receiving antidepressant, antianxiety, antipsychotic, or mood-stabilizer medication where the dose has not been stable for a minimum of six weeks prior to entering the randomization
6. evidence of receiving psychosocial or medication treatment through a clinic or facility other than the VA GLA PTSD Clinic.
7. infection or loss of integrity of skin over the forehead, where the electrode pads will be placed.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VA PTSD Clinic, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at the VA Greater Los Angeles and VA Long Beach.
Pre-assignment Details: 95 Potential participants were assessed for eligibility, of the 95, 23 participants did not meet the study criteria, and 72 participants were consented for the study.
  Of the 72 consented participants, 12 subjects dropped prior to randomization resulting in 60 randomized, evaluable participants.
Groups:
- Sham: The stimulators are the same device for the active and sham treatment conditions.
  Placebo: Subjects will be randomized to treatment with either active or sham Trigeminal Nerve Stimulation (TNS) for a period of eight weeks. The programming will be set by an individual who has no contact with subjects to deliver TNS in a double-blind manner (n=37 in each group) at the sham frequency of 0 Hz. TNS will be performed for approximately 8 hours each night, a protocol that subjects found acceptable in the pilot work.
- Active: The stimulators are the same device for the active and sham treatment conditions.
  Trigeminal Nerve Stimulation (TNS): Subjects will be randomized to treatment with either active or sham TNS for a period of eight weeks. The programming will be set by an individual who has no contact with subjects to deliver TNS in a double-blind manner (n=37 in each group) at the active frequency of 120 Hz. TNS will be performed for approximately 8 hours each night, a protocol that subjects found acceptable in the pilot work.
Period: Overall Study
Arm/Group | Sham | Active
Started | 31 | 29
Completed | 22 | 24
Not Completed | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham | Active | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 29 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 41.33 [26 to 55] | 35.57 [19 to 50] | 37.71 [19 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 31 | 27 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Treatment Efficacy as Measured by Change in Clinician-Administered Post Traumatic Stress Disorder Score for Diagnostic and Statistical Manual of Mental Disorders, 5th Edition(DSM-V) at Baseline and Week 8 Visit
Description: Treatment efficacy as measured by change in Clinician-Administered Post Traumatic Stress Disorder score for Diagnostic and Statistical Manual of Mental Disorders, 5th Edition at baseline and Week 8 visit. This is a 30-item questionnaire with minimum and maximum score values ranging from 0 to 80. Higher scores indicate a worse outcome and lower scores indicate better outcome.
Time Frame: 8 weeks (Baseline visit and Week 8 visit)
Population: Discrepancy in subjects randomized and subjects analyzed reflect the number of subjects who were randomized but discontinued intervention prior to reaching an evaluable time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Sham: The stimulators are the same device for the active and sham treatment conditions.
  Placebo: Subjects will be randomized to treatment with either active or sham TNS for a period of eight weeks. The programming will be set by an individual who has no contact with subjects to deliver TNS in a double-blind manner (n=31 in sham group) at the sham frequency of 0 Hz. TNS will be performed for approximately 8 hours each night, a protocol that subjects found acceptable in the pilot work.
- Active: The stimulators are the same device for the active and sham treatment conditions.
  Trigeminal Nerve Stimulation: Subjects will be randomized to treatment with either active or sham TNS for a period of eight weeks. The programming will be set by an individual who has no contact with subjects to deliver TNS in a double-blind manner (n=29 in active group) at the active frequency of 120 Hz. TNS will be performed for approximately 8 hours each night, a protocol that subjects found acceptable in the pilot work.
Arm/Group | Sham | Active
Number analyzed (Participants) | 26 | 28
score on a scale
  Baseline | 50.60 (6.83) | 50.10 (7.77)
  Week 8 | 28.29 (14.74) | 28.61 (12.99)

2. Secondary Outcome: Treatment Efficacy as Measured by Change in Score on Beck Depression Inventory-II Assessment Scores.
Description: Secondary outcome measures will be the change in Beck Depression Inventory-II scores from Baseline to Week 8. This is a 21-item scale with maximum and minimum scores ranging from 0 to 63. Higher scores indicate a worse outcome and lower scores indicate a better outcome. For examination of change scores, baseline represents the scores at the time of the second baseline visit (immediately prior to the start of treatment). The endpoint for comparison to baseline will be the week 8 time point or the last non-missing observation during the double-blind treatment.
Time Frame: 8 weeks ((Baseline visit and Week 8 visit)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham | Active
Number analyzed (Participants) | 26 | 28
score on a scale
  Baseline | 28.29 (9.41) | 28.31 (9.43)
  Week 8 | 15.36 (9.28) | 15.78 (12.55)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected each weekly assessment visit for every participant, up to 8 weeks
Description: Serious Adverse events remain at zero as the research treatment administered in this study is categorized as minimal risk and non-significant risk. This indicates an inherent lack of risk for death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, a congenital anomaly/birth defect, or all-cause mortality.
Arm/Group | Sham | Active
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 0/31 | 1/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham (N=31) | Active (N=29)
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Treatment emergent headaches described as mild to moderate were reported by one participant. Subject discontinued participation due to this event. Headaches did not persist after discontinuation of use. This is an anticipated adverse event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT02377089/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT02377089/ICF_001.pdf